CLINICAL TRIAL: NCT02747862
Title: Non-Surgical Management of Attenuated and Deleterious (Classical) Familial Adenomatous Polyposis: A Long-term Surveillance Program
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: DR08-0006
Record Dates: First submitted 2016-04-14; First posted 2016-04-22 (Estimated); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Attenuated Familial Adenomatous Polyposis; Deleterious Familial Adenomatous Polyposis
Keywords: Attenuated Familial Adenomatous Polyposis; AFAP; Deleterious Familial Adenomatous Polyposis; FAP; Chart review
MeSH Terms: conditions — Attenuated familial adenomatous polyposis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Attenuated Familial Adenomatous Polyposis: Chart review study to evaluate the outcomes of subjects with Attenuated Familial Adenomatous Polyposis (AFAP) who have not undergone surgical resection of the colon.
  Interventions: Other: Chart Review
- Deleterious Familial Adenomatous Polyposis: Chart review study to evaluate the outcomes of subjects with Deleterious Familial Adenomatous Polyposis (FAP) who have not undergone surgical resection of the colon.
  Interventions: Other: Chart Review

INTERVENTIONS:
Other: Chart Review — Database queried for the presence of cases meeting criteria (attenuated FAP, classical AFP [i.e. identifiable APC mutation], and/or a compatible family history or personal adenoma burden of > 50 adenomas).
  The data related to the patients with attenuated FAP and classical AFP who underwent endoscopic surveillance or surgery collected through chart review and all data is retrospective as of February 15, 2016.

SUMMARY:
The primary objective of this chart review study is to evaluate the outcomes of subjects with Attenuated Familial Adenomatous Polyposis (AFAP) and Deleterious Familial Adenomatous Polyposis (FAP) who have not undergone surgical resection of the colon.

A secondary objective of this study is to compare 1) the colonoscopic and pathology histories including history of ampullary adenoma in the duodenum over family generations, 2) the use of chemopreventive medications, and 3) clinical features of subjects who pursued prophylactic surgical resection of the colon with those that have elected to continue routine colonoscopic surveillance in an effort to better characterize factors (e.g. polyp burden, ampullary adenoma and level of dysplasia, etc) which may influence management decisions.

DETAILED DESCRIPTION:
The UTMDACC family history database will be queried for the presence of cases meeting the above criteria (attenuated Familial Adenomatous Polyposis (FAP), classical AFP [i.e. identifiable APC mutation], and/or a compatible family history or personal adenoma burden of > 50 adenomas).

The data related to the patients with attenuated FAP and classical AFP who underwent endoscopic surveillance or surgery will be collected through chart review and all data is retrospective as of February 15, 2016.

The University of Texas MD Anderson Cancer Center (UTMDACC) medical record number for these cases will be used to identify the patient in ClinicStation: 1) records of endoscopy procedures, 2) operative reports, and 3) associated clinic notes will be reviewed for: a) whether the above evaluation criteria have been met, b) age, c) gender, d) age at initial colonoscopy, e) total number of colonoscopies, f) number of adenomas identified, g) cancer diagnoses, h) chemopreventive medications, i) type of surgery, j) number of hospitalizations, k) length of hospital stay, l) identification of an underlying APC mutation, and ll) family history information. The UT MDACC family history database will also be reviewed for updated family history information including ampullary adenomas and outcomes of genetic testing for identified cases.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with either a genetic diagnosis of AFAP/FAP (i.e. an identifiable APC gene mutation), and/or a compatible family history and pathology including history of ampullary adenoma in the duodenum over family generations, or personal adenoma burden of > 50 adenomas are to be included.

Exclusion Criteria:

1. Participants who do not have with Attenuated Familial Adenomatous Polyposis (AFAP) and Deleterious Familial Adenomatous Polyposis (FAP).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants with either a genetic diagnosis of AFAP/FAP (i.e. an identifiable APC gene mutation), and/or a compatible family history and pathology including history of ampullary adenoma in the duodenum over family generations, or personal adenoma burden of > 50 adenomas at MD Anderson Cancer Center in Houston, Texas.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2008-02 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2022-08-17 (Actual)

PRIMARY OUTCOMES:
Chart Review of Outcomes of Participants with Attenuated Familial Adenomatous Polyposis (AFAP) and Deleterious Familial Adenomatous Polyposis (FAP) Undergoing Endoscopic Surveillance | 12 years
  For comparisons between groups, the Mann-Whitney test used.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Lynch, MD, JD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org